CLINICAL TRIAL: NCT03713853
Title: GATOR: Geriatric Acetabular fracTures: Open Reduction Internal Fixation Versus Replacement - A Large Cohort of Acute Open Reduction Internal Fixation (ORIF) Versus Total Hip Arthroplasty for Geriatric Acetabular Fractures
Brief Title: Geriatric Acetabular fracTures: Open Reduction Internal Fixation Versus Replacement
Acronym: GATOR
Status: Recruiting | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 18-0303
Record Dates: First submitted 2018-10-16; First posted 2018-10-22 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Acetabular Fracture
Keywords: Total hip replacement; Total hip arthroplasty; Open Reduction internal Fixation; Hip fixation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Total hip arthroplasty + ORIF: Patients will receive acute primary total hip arthroplasty (THA) with open reduction internal fixation (ORIF) as a treatment for their acetabular fracture
- Surgical Fixation (ORIF): Patients will receive open reduction internal fixation (ORIF) as a treatment for their acetabular fracture

SUMMARY:
Management of acetabular (hip) fractures in the geriatric population can be very challenging because of pre-existing medical comorbidities, pre-existing osteoporosis and increased risk of mortality.

The two most common treatment options for acetabular fractures are either surgical fixation using plates and screws to hold the fractured pieces in the correct position until the fracture has healed or surgical fixation in addition to a total hip replacement.

Surgical fixation requires prolonged immobilization of the affected limb (typically around 6-12 weeks post-operatively), which can lead to disability and other complications. Such patients, especially those who are frail and cognitively impaired, are unable to adhere to the immobilization restrictions, leading to an increased risk of fixation failure.

Patients who underwent open reduction internal fixation (ORIF) of an acetabular fracture were reported to have about 25 times greater incidence of hip replacement compared with general population matched controls.

Additionally, performing a subsequent hip replacement after a previous surgical fixation (ORIF) of an acetabular fracture, especially in the elderly population, can present a number of technical difficulties including; difficult dissection due to previous incision(s) and scarring, dealing with retained hardware, bony deficiency and the possibility of infected hardware.

The aim of the study is to perform a large cohort study to assess pain and physical function in patients 60 years and older who have sustained an acetabular fracture.

DETAILED DESCRIPTION:
This is a multicentre observational cohort study, involving academic institutions affiliated with the Canadian Orthopaedic Trauma Society (COTS).

The study aims to compare two surgical treatments of acetabular fractures in patients 60 years of age and older. Patients who consent to participate will be included in the study and followed up as per standard of care up to 24 months after surgery. Participants will be treated for their acetabular fracture with either acute primary total hip arthroplasty (THA) together with open reduction internal fixation (ORIF) in the same surgery or ORIF alone as per surgeon discretion.

After surgery, patients will be assessed using patient-reported outcomes oxford hip score, which is a valid, reliable, responsive measure of pain and function during short-term and long-term follow-up for hip osteoarthritis and THA.

The European Quality of Life-5 Dimensions (EQ-5D), will be used to assess the patient's quality of life and health status. The questionnaire is short and easy to use and shows good responsiveness in orthopaedic patients who undergo a hip replacement.

Timed Up & Go Test (TUG) measures functional mobility (in seconds), and is a well-validated predictor of mobility and falls in patients who undergo orthopaedic surgery and hip replacement.

All patients will be followed as per standard of care for their follow up visits at 6 weeks, 3, 6, 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older
* Isolated and Displaced (more or equal to 2mm on any radiographic view) fracture of the acetabulum
* Patient requires surgical treatment, either THA+ORIF or ORIF surgeries
* Fracture is acute (within 3 weeks of injury)
* Patient was ambulatory (with or without walking aids) prior to their acetabular fracture injury
* Patient is able to provide informed consent to participation in the study
* Patient is able to read and understand English

Exclusion Criteria:

* Presence of an active or chronic infection around the fracture (soft tissue or bone)
* Open/compound fracture
* Bilateral acetabular fractures
* Pathological fracture excluding osteoporosis
* Periprosthetic fracture (previous arthroplasty or hardware or ORIF in-situ). Hardware (screws or plates or nails or hemi-arthroplasty) on the femoral side are not excluded.
* Medical or surgical contraindication to surgery
* Dementia

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients 60 years of age and older, presenting at the participant hospital sites with a displaced acetabular fracture and who need surgery to fix their fracture, either total hip replacement (THA) together with surgical fixation (ORIF) or surgical fixation (ORIF) alone, will be screened for the study.
  Patients who meet the trial eligibility criteria will be approached by a member of the research team. The study will be explained in detail and written informed consent will be undertaken with those patients who wish to participate in the study. Outcomes for participants will be measured and captured during regularly scheduled clinic/hospital visits
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Oxford Hip score | Questionnaire will be completed by patients at 3, 6 and 12-months follow-up and repeated measures analysis will be performed to assess the change across all time points (3,6 and 12-months)
  Oxford Hip Score is a short 12-item patient-reported outcome specifically designed and developed to assess function and pain during short-term and long-term follow-up for hip osteoarthritis and hip replacement surgery. It is valid, reliable, reproducible, and sensitive to clinically important changes. An increase in score indicate better joint function. A score between 40-48 indicates satisfactory joint function.

SECONDARY OUTCOMES:
Timed Up and Go (TUG) test | Test will be completed at 3, 6,12 and 24-months follow-up
  TUG is a simple test used to assess a person's mobility (in seconds) and requires both static and dynamic balance. A line is placed on the floor 3 meters away from a chair where patient will be sitting.
  When instructed to "GO" patient will stand, walk to a line on the floor at his/her regular pace, turn around and walk back to the chair and sit down.
  The longer it takes for subject to complete the test, higher is the risk of fall and lower is the its functional mobility.
  Reference values are:
  60-69 years old = 8.1 seconds; 70-79 years old = 9.2 seconds; 80-99 years old = 11.3 seconds. Over 14 seconds is associate with high risk of fall
Visual Analogue Scale of pain (VAS) | Patients will indicate their pain level at 24, 48 hours, 6 weeks, 3, 6,12 and 24-months after surgery
  Assess pain from a visual scale that ranges from 0 to 10. Straight line with the endpoints defining extreme limits such as 'no pain at all' (zero) and 'pain as bad as it could be' (ten)
Total Morphine Equivalents Usage | The outcome will be assessed daily from the day of the surgery until the patient gets discharge from the hospital (24 hours up to 7 days)
  The sum (cumulative) of amount of opiates dosage (in milligram) prescribed daily (24hours) and converted in total morphine equivalent dosage (total dosage every 24 hours).
Health status and quality of life | Questionnaire will be completed by patients at 6 weeks, 3, 6, 12 and 24-months follow-up
  The European Quality of Life-5 Dimensions (EQ-5D) is a patient-reported outcome where patients self-rate their level of severity of health status and health related quality of life. Consists of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and each one of them has 5 levels (no problems, slight problems, moderate problems, severe problems, and extreme problems) where patients will indicate how they feel regarding their health status and quality of life.
Length of hospital stay | The outcome will be assessed from the day of the surgery until the patient gets discharge from the hospital (at a maximum of 30 days after the surgery)
  How many days the patient stay in the hospital
Discharge location | from the day of the surgery until the patient gets discharge from the hospital
  Site where the patient gets discharge, such as home, rehabilitation, acute care facility
Time to full-weight bearing | Since the first day after surgery up to 12 months
  time (in days) that takes for the patient to start walking after the surgery
Time to return to work and activities of daily life | from the day of the surgery up to 24 months follow up
  How many days until the patients return to their normal daily life activities such as independently walking, bathing/showering, grooming, dressing, etc. and How many days until patients return to work
Hospital Re-admission | Within 30 days of discharge
  Any admission to any hospital after the patients is discharge from the hospital where he/she underwent the surgical treatment for acetabular fracture

CONTACTS AND LOCATIONS:
Overall Officials: Amir Khoshbin, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- Unity Health Toronto - St Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cahueque M, Martinez M, Cobar A, Bregni M. Early reduction of acetabular fractures decreases the risk of post-traumatic hip osteoarthritis? J Clin Orthop Trauma. 2017 Oct-Dec;8(4):320-326. doi: 10.1016/j.jcot.2017.01.001. Epub 2017 Jan 13. PMID 29062212
- [Background] Firoozabadi R, Cross WW, Krieg JC, Routt MLC. Acetabular Fractures in the Senior Population- Epidemiology, Mortality and Treatments. Arch Bone Jt Surg. 2017 Mar;5(2):96-102. PMID 28497099
- [Background] Boelch SP, Jordan MC, Meffert RH, Jansen H. Comparison of open reduction and internal fixation and primary total hip replacement for osteoporotic acetabular fractures: a retrospective clinical study. Int Orthop. 2017 Sep;41(9):1831-1837. doi: 10.1007/s00264-016-3260-x. Epub 2016 Aug 10. PMID 27511470
- [Background] Hanschen M, Pesch S, Huber-Wagner S, Biberthaler P. Management of acetabular fractures in the geriatric patient. SICOT J. 2017;3:37. doi: 10.1051/sicotj/2017026. Epub 2017 May 25. PMID 28534471
- [Background] Morison Z, Moojen DJ, Nauth A, Hall J, McKee MD, Waddell JP, Schemitsch EH. Total Hip Arthroplasty After Acetabular Fracture Is Associated With Lower Survivorship and More Complications. Clin Orthop Relat Res. 2016 Feb;474(2):392-8. doi: 10.1007/s11999-015-4509-1. PMID 26335343
- [Background] Khurana S, Nobel TB, Merkow JS, Walsh M, Egol KA. Total Hip Arthroplasty for Posttraumatic Osteoarthritis of the Hip Fares Worse Than THA for Primary Osteoarthritis. Am J Orthop (Belle Mead NJ). 2015 Jul;44(7):321-5. PMID 26161760
- [Background] Henry PDG, Si-Hyeong Park S, Paterson JM, Kreder HJ, Jenkinson R, Wasserstein D. Risk of Hip Arthroplasty After Open Reduction Internal Fixation of a Fracture of the Acetabulum: A Matched Cohort Study. J Orthop Trauma. 2018 Mar;32(3):134-140. doi: 10.1097/BOT.0000000000001048. PMID 29462122
- [Background] O'Toole RV, Hui E, Chandra A, Nascone JW. How often does open reduction and internal fixation of geriatric acetabular fractures lead to hip arthroplasty? J Orthop Trauma. 2014 Mar;28(3):148-53. doi: 10.1097/BOT.0b013e31829c739a. PMID 23719343
- [Background] Weaver MJ, Smith RM, Lhowe DW, Vrahas MS. Does Total Hip Arthroplasty Reduce the Risk of Secondary Surgery Following the Treatment of Displaced Acetabular Fractures in the Elderly Compared to Open Reduction Internal Fixation? A Pilot Study. J Orthop Trauma. 2018 Feb;32 Suppl 1:S40-S45. doi: 10.1097/BOT.0000000000001088. PMID 29373451
- [Background] Hamlin K, Lazaraviciute G, Koullouros M, Chouari T, Stevenson IM, Hamilton SW. Should Total Hip Arthroplasty be Performed Acutely in the Treatment of Acetabular Fractures in Elderly or Used as a Salvage Procedure Only? Indian J Orthop. 2017 Jul-Aug;51(4):421-433. doi: 10.4103/ortho.IJOrtho_138_16. PMID 28790471
- [Background] Ortega-Briones A, Smith S, Rickman M. Acetabular Fractures in the Elderly: Midterm Outcomes of Column Stabilisation and Primary Arthroplasty. Biomed Res Int. 2017;2017:4651518. doi: 10.1155/2017/4651518. Epub 2017 Jan 17. PMID 28194414